CLINICAL TRIAL: NCT02680730
Title: The Listening Project at the ADD Centre and Biofeedback Institute of Toronto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: ADD Centre© and Biofeedback Institute of Toronto© (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-1954
Record Dates: First submitted 2016-02-08; First posted 2016-02-11 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Auditory Perceptual Disorders; Stress Disorder
Keywords: Autonomic nervous system; Auditory processing disorder; Social behavior
MeSH Terms: conditions — Auditory Perceptual Disorders; Stress Disorders, Traumatic; Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention only (Experimental): Participants will be included in 1 pre-intervention and 2 post-assessment measures. Participants will receive the Listening Project Protocol intervention (filtered music). The duration of the intervention is approximately 60 minutes per day, for 5 consecutive days.
  Interventions: Behavioral: Listening Project Protocol
- Intervention + Stability (Experimental): Participants will be included in 2 pre-intervention and 2 post-assessment measures. The additional pre-intervention assessment will allow for assessment of stability of measures. Participants will receive the Listening Project Protocol intervention (filtered music). The duration of the intervention is approximately 60 minutes per day, for 5 consecutive days.
  Interventions: Behavioral: Listening Project Protocol

INTERVENTIONS:
Behavioral: Listening Project Protocol — The filtered-music intervention will consist of listening to computer-altered acoustic stimulation, designed to modulate the frequency band of vocal music passed to the participant. The frequency characteristics of the acoustic stimulation are selected to emphasize the relative importance of specific frequencies in conveying the information embedded in human speech. Modulation of the acoustic energy within the frequencies of human voice, similar to an exaggerated vocal prosody, are hypothesized to recruit and modulate the neural regulation of the middle ear muscles and to functionally reduce sound hypersensitivities and improve auditory processing.

SUMMARY:
Purpose: A research project will be conducted at the ADD ("Attention Deficit Disorder") Centre and Biofeedback Institute of Toronto to evaluate the feasibility of the Listening Project Protocol (LPP) intervention in individuals with difficulties with autonomic and/or behavioral regulation. The LPP is designed as a "neural exercise" to reduce auditory hypersensitivities, to improve auditory processing of speech, and to improve behavioral state regulation. These improvements should translate into increase feelings of safety and calmness, thereby promoting improvement in social behavior.

Participants: 30 participants, males and females between ages 7-55 years, will be recruited for the study. Participants will be patients at the ADD Centre and Biofeedback Institute of Toronto.

Procedures: Participants will be divided into 1 of 2 groups (1:1 ratio). Both groups will have a pre-intervention assessment #2, intervention, 1 week post intervention assessment and 1 month post intervention assessment. Group 2 will have an additional pre-intervention assessment session #1 (1 week previous to pre-intervention assessment #2) to assess the stability of the measures prior to starting the intervention. Pre-, post-, and 1 month followup assessment will include parent and/or self-report questionnaires, and measures of the individual's auditory processing ("SCAN"), affect recognition ("DARE" Dynamic Affect Recognition Evaluation), heart rate, prosody, "RSA" respiratory sinus arrhythmia (derived from non-invasive ECG recording), and middle ear transfer function ("MESAS" - Middle Ear Sound Absorption System).

ELIGIBILITY:
Inclusion Criteria:

1. Individuals must be between ages 7-55 years
2. Individuals must be fluent (read and write) in English. Parents must be able to read/speak in English.
3. Individuals must be current or past clients at the ADD Centres Limited & Biofeedback Institute of Toronto

Exclusion criteria:

1. Individuals who wear a hearing-device
2. Individuals with a history of heart disease
3. Individuals who are currently being treated for seizure disorder
4. Individuals who are non-verbal

Ages: 7 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in auditory hypersensitivity at 1 week, and at 1 month | pre-intervention (within 1 week before intervention), post-intervention (within 1 week after intervention), 1 month post-intervention
  Brain-Body Center Sensory Scales (BBC Sensory Scales) (parental questionnaire)

SECONDARY OUTCOMES:
Change from baseline in state regulation at 1 week, and at 1 month | pre-intervention (within 1 week before intervention), post-intervention (within 1 week after intervention), 1 month post-intervention
  heart rate, heart period, high-frequency heart rate variability/respiratory sinus arrhythmia
Change from baseline in auditory processing at 1 week, and at 1 month | pre-intervention (within 1 week before intervention), post-intervention (within 1 week after intervention), 1 month post-intervention
  filtered words, competing words subscales of SCAN-3:C Tests for Auditory Processing Processing Disorders in Children
Change from baseline in social behavior at 1 week, and at 1 month | post-intervention (within 1 week after the intervention), 1 month post-intervention
  Listening Project Parent Questionnaire
Change from baseline in middle ear transfer function at 1 week, and at 1 month | pre-intervention (within 1 week before intervention), immediate post-intervention (within 1 week after intervention), 1 month post-intervention
  Middle Ear Sound Absorption System (MESAS)
Change from baseline in prosody at 1 week, and at 2 months | pre-intervention (within 1 week before intervention), immediate post-intervention (within 1 week after intervention), 1 month post-intervention
  Prosody assessment of recorded speech
Change from baseline in attention at 1 week, and at 2 months | pre-intervention (within 1 week before intervention), immediate post-intervention (within 1 week after intervention), 1 month post-intervention
  Connors Questionnaire
Change from baseline in attention (task) at 1 week, and at 2 months | pre-intervention (within 1 week before intervention), immediate post-intervention (within 1 week after intervention), 1 month post-intervention
  Integrated Visual and Auditory Continuous Performance Task ("IVA")

CONTACTS AND LOCATIONS:
Overall Officials: Keri J Heilman, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- ADD Centre and Biofeedback Institute of Toronto, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No